CLINICAL TRIAL: NCT00426400
Title: Anti-Aggregative Therapy and Laser Iridectomy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHEBA-05-3876-HLV-CTIL
Record Dates: First submitted 2006-10-25; First posted 2007-01-24 (Estimated); Last update posted 2007-01-24 (Estimated); Status verified 2007-01

CONDITIONS: Eyes With Narrow Angle

INTERVENTIONS:
Drug: The cessation of anti-aggregative treatment for 10 days

SUMMARY:
Our study investigates the effect of anti-aggregative treatment on success and complications of laser iridectomy. The study includes patients scheduled for laser iridectomy due to narrow angles.Patients will undergo first laser treatment with the anti-aggregative treatment and will scheduled for next lase in the other eye after discontinuing the anti-aggregative treatment. The patients will be followed-up for 3 months.

ELIGIBILITY:
Inclusion Criteria:

* patients with narrow angle that need laser iridectomy and take anti- aggregative treatment
* over 20 years old
* patients who can stop their anti-aggregative treatment for 10 days

Exclusion Criteria:

* under coumadin treatment
* post ocular surgeries

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2006-03

CONTACTS AND LOCATIONS:
Overall Officials: Hani Levkovitch-Verbin, MD, Principal Investigator — Goldscheleger Eye Institute, Sheba Medical Center
Locations (1):
- Goldschleger Eye Institute, Tel Litwinsky, Israel